CLINICAL TRIAL: NCT05519423
Title: Investigation of the Effectiveness of Whatsapp-Based Physical Activity Incentive Program in Morbidly Obese Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gulfidan Tokgoz, Lecturer, PT, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022/241
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Physical Inactivity; Obesity, Morbid
Keywords: physical activity; morbid obesity; exercise; technology
MeSH Terms: conditions — Sedentary Behavior; Obesity, Morbid; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Morbid obesity individuals (Experimental): All subjects participating in the study will be given physical activity incentive program (PAI) individually. After evaluating it is aimed to provide information transfer and motivation support to increase physical activity levels before bariatric surgery within the scope of PAI.
  For this purpose, individual face-to-face interviews will conduct with all cases; verbal information will be given about the importance of physical activity, its effects and different levels of severity. The progress of the program will be made with the whats app application.
  8-week follow-up chart will be given to the individuals, about the completion of the physical activity follow-up chart prepared in order to raise awareness about the activity levels of individuals in daily life and to increase their physical activity levels.
  All subjects will record daily step counts, low, moderate, and vigorous activities on the chart at the end of the day, every day for 8 weeks.
  Interventions: Behavioral: Physical Activity Incentive Program

INTERVENTIONS:
Behavioral: Physical Activity Incentive Program — Physical Activity Incentive (PAI) programs, which is a method used in preventive health services, are recommended by a number of public health institutions, including the World Health Organization, thanks to the universal access and high potential of health services. PAI is defined as offering verbal or written advice/guidance to encourage the individual to increase their current level of physical activity.

SUMMARY:
The limited number of studies on the effectiveness of physical activity incentive programs for morbidly obese individuals in the literature shows the need in this area.

In this study, primary aim is to investigate the effect of physical activity incentive program applied through face-to-face and whatsapp-based applications on physical activity level, functional capacity and muscular endurance in morbidly obese individuals.

Secondary aim is to provide individuals with exercise habits and to ensure participants' sustainability with the physical activity incentive program planned in line with the needs of the individual.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 18-60
* BMI ≥40 kg/m2, morbidly obese awaiting bariatric surgery
* No surgical operation in the last 6 months

Exclusion Criteria:

* Having a musculoskeletal disorder or systemic disease that will interfere with physical activity
* Presence of balance problems that will prevent physical activity
* Presence of psychiatric or neurological disease affecting cooperation and cognitive functions
* Presence of acute pain
* Heartache
* Having a history of myocardial infarction
* Presence of conjunctive heart failure
* Presence of uncontrolled diabetes and hypertension

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
The International Physical Activity Questionnaires (IPAQ) | up to 8 weeks
  The short form of the International Physical Activity Questionnaire (IPAQ) will be used to determine the physical activity levels of the participants. The IPAQ-Short Form is a valid tool used to assess physical activity in young adults. It is a 7-item scale that evaluates the duration and frequency of vigorous physical activity, moderate physical activity, walking and sedentary behavior based on MET values. Physical activity levels are classified into 3 categories according to the scores obtained by multiplying the duration, frequency and MET values of the physical activities that the participants participated in within 7 days and for at least 10 minutes. Accordingly, <600 MET - min/week is defined as inactive, 600 - 3000 MET - min/week low, and >3000 MET - min/week is defined as sufficient physical activity level.

SECONDARY OUTCOMES:
Bioelectrical Impedance Analysis (BIA) Measurement | up to 8 weeks
  The muscle, fat, and water ratio of the cases were evaluated with the Inbody Bioelectrical Impedance Device.
6 Minute Walk Test | up to 8 weeks
  According to the guide published by the American Thoracic Society, the 6MWT is easy to administer, better tolerated, and better reflecting daily activities than other walking tests. It can be applied in a short time in a limited space and requires little equipment. 6MWT is used in various disease groups to evaluate functional capacity.
Sit and Stand Test | up to 8 weeks
  In order to evaluate the muscular endurance of the subjects, the participant sitting in a 43 cm high standard chair with his arms crossed over his shoulders is asked to stand up and sit down quickly for 30 seconds, and the number of repetitions at which full rise is achieved will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Gulfıdan Tokgoz, Principal Investigator — İstanbul University-Cerrahpasa; Nilay Arman, Principal Investigator — İstanbul University-Cerrahpasa; Hakan Seyit, Principal Investigator — BAKIRKOY DR. SADİ KONUK EDUCATION AND RESEARCH HOSPITAL; Mehmet Karabulut, Principal Investigator — BAKIRKOY DR. SADİ KONUK EDUCATION AND RESEARCH HOSPITAL
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Physical Activity Strategy for the WHO European Region 2016-2025; World Health Organisation Regional Office for Europe: Copenhagen, Denmark, 2016; ISBN 9289051477.
- [Background] van Poppel MN, Chinapaw MJ, Mokkink LB, van Mechelen W, Terwee CB. Physical activity questionnaires for adults: a systematic review of measurement properties. Sports Med. 2010 Jul 1;40(7):565-600. doi: 10.2165/11531930-000000000-00000. PMID 20545381
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Solway S, Brooks D, Lacasse Y, Thomas S. A qualitative systematic overview of the measurement properties of functional walk tests used in the cardiorespiratory domain. Chest. 2001 Jan;119(1):256-70. doi: 10.1378/chest.119.1.256. PMID 11157613